CLINICAL TRIAL: NCT01058109
Title: Effect of Calcium Foods on Bone Quality in Pubertal Females
Brief Title: Study of the Effect of a Calcium-rich Diet on Bone Health in Girls
Acronym: Calkids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Joan Lappe, Professor of Medicine, Creighton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 97-11179
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Bone Health
Keywords: bone health, bone density, bone mass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- calcium group (Experimental): dietary calcium intake of 1500 mg/d
  Interventions: Other: calcium-rich diet
- calcium-rich diet (1500 mg/d) (Experimental): calcium intake from food
  Interventions: Other: Calcium rich diet

INTERVENTIONS:
Other: calcium-rich diet — dietary calcium intake of 1500 mg/d
  Arms: calcium group
Other: Calcium rich diet — dietary intake of 1500 mg/d from food
  Arms: calcium-rich diet (1500 mg/d)

SUMMARY:
The aim of this experimental study was to test the effect of increasing dietary calcium intake to 1500 mg/day on increases in bone quality in adolescent females. The hypothesis to be tested is: adolescent females who consume a high calcium diet will have a greater increase in bone quality, as measured by densitometry and ultrasound, than adolescent females who consume their usual dietary calcium intake.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria were being female and nine years of age with usual dietary calcium intake 1100 mg/day or less.

Exclusion Criteria:

* Exclusion criteria included history of any of the following: lactose intolerance, milk allergy, corticosteroid or anticonvulsant therapy, familial hypercholesterolemia, mental or physical handicaps, cancer, rheumatoid arthritis, asthma, or any significant health problem reported by the parents. We also excluded any child who had a body mass index (BMI)85th percentile for age and gender and children who practiced or played any organized sport (including gymnastics or dance) more than three times per week.

Ages: 9 Years to 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 1997-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The specific aim of this project was to test the effect of increasing dietary calcium intake to 1500 mg/day on increases in bone quality in pubertal females beginning at age nine. | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Lappe, PhD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States